CLINICAL TRIAL: NCT05150548
Title: Development and Internal Validation of Models to Predict Time-to-event for Major Medical Complications Within 30-days After Planned Colectomy: a Retrospective Population Cohort Study
Brief Title: Predictive Time-to-Event Model for Major Medical Complications After Colectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Janny Ke, Clinical Instructor, University of British Columbia
Other Study IDs: H21-02670
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer; Inflammatory Bowel Diseases; Diverticulitis; Colectomy; Predictive Model; Complications, Postoperative
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases; Diverticulitis; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Entire Cohort: Patients undergoing elective colectomy with data that has been collected in the NSQIP® Procedure Targeted Colectomy dataset from 2014-2019 with American Society of Anesthesiologists (ASA) Physical Status I-IV.
  Patients will not be included in this cohort with urgent or emergency colectomy or indication for colectomy consisting of "Acute diverticulitis", "Enterocolitis (e.g. C. Difficile)", and "Volvulus", patients with disseminated cancer, wound infection, systemic sepsis or ventilator-dependence preoperatively.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Not applicable, non-interventional study

SUMMARY:
Purpose: The purpose of this study is to create prediction models for when major complications occur after elective colectomy surgery.

Justification: After surgery, patients can have multiple complications. Accurate risk prediction after surgery is important for determining an appropriate level of monitoring and facilitating patient recovery at home.

Objectives: Investigators aim to develop and internally validate prediction models to predict time-to-complication for each individual major medical complications (pneumonia, myocardial infarction (MI) (i.e. heart attacks), cerebral vascular event (CVA) (i.e. stroke), venous thromboembolism (VTE) (i.e. clots), acute renal failure (ARF) (i.e. kidney failure), and sepsis (i.e. severe infections)) or adverse outcomes (mortality, readmission) within 30-days after elective colectomy.

Data analysis: Investigators will be analyzing a data set provided by the National Surgical Quality Improvement Program (NSQIP). Descriptive statistics will be performed. Cox proportional hazard and machine learning models will be created for each complication and outcome outlined in "Objectives". The performances of the models will be assessed and compared to each other.

DETAILED DESCRIPTION:
Background: Planned (elective or time sensitive) colectomy are performed for indications including cancer, inflammatory bowel disease (IBD), and diverticulitis. After colectomy, patients are at risk of a variety of major medical complications, including pneumonia, myocardial infarction (MI), cerebral vascular event (CVA), venous thromboembolism (VTE), acute renal failure (ARF), and sepsis. However, different complications tend to happen at different times after surgery. Accurate risk prediction, not only whether a complication may occur in a patient, but also when, is crucial for patient education, monitoring, and disposition planning. While several studies have explored the incidence and binary risk prediction for major complications after surgeries, there has been scarce literature on time-to-complication prediction modeling in recent population cohort data.

Objectives

1. To develop and internally validate Cox proportional hazards models to predict time-to-complication for each individual major medical complication captured in the American College of Surgeons National Surgical Quality Improvement Program (NSQIP) dataset (pneumonia, myocardial infarction (MI), cerebral vascular event (CVA), venous thromboembolism (VTE), acute renal failure (ARF), and sepsis) or adverse outcomes (mortality, readmission), that started within 30-days after elective colectomy.
2. To develop and internally validate machine learning models to predict time-to-complication for major medical complications and adverse outcomes (same as in objective 1) within 30-days after elective colectomy in NSQIP. The best machine learning model for each complication will be compared to the Cox proportional hazards model in terms of discrimination, and calibration.

Methods: Investigators will conduct a time-to-event survival analysis in a retrospective cohort using NSQIP®, a prospectively-collected multicentre dataset with more than 150 clinical variables within 30 days after surgery. This dataset includes information on whether the patient was diagnosed with major complications (in- or out-of-hospital) as well as the number of postoperative days to the diagnoses of complications, as defined by a standardized criteria within the NSQIP operations manual. The general dataset will be linked with the NSQIP® Procedure Targeted Colectomy dataset, which contains additional colectomy-specific variables.

The study will be reported according to the Transparent reporting of a multivariable prediction model for individual prognosis or diagnosis (TRIPOD) guidelines and Guidelines for Developing and Reporting Machine Learning Predictive Models in Biomedical Research.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective colectomy
* data has been collected in the NSQIP® Procedure Targeted Colectomy dataset from 2014-2019

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status (PS) V (defined as "5-Moribund") (ASA PS 6 - organ donation is not included within NSQIP)
* undergoing urgent or emergency surgery
* indication for colectomy consisting of "Acute diverticulitis", "Enterocolitis (e.g. C. Difficile)", and "Volvulus" due to the non-elective nature of these pathologies
* patient with disseminated cancer
* wound infection (i.e. potentially recent surgery)
* systemic sepsis
* ventilator-dependence preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include all patients who are 18 years or older undergoing elective colectomy, whose data has been collected in the NSQIP® Procedure Targeted Colectomy dataset from 2014-2019, inclusively.
Sampling Method: Probability Sample
Enrollment: 130000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pneumonia | Within 30 days post-operatively
  Occurrence of pneumonia within 30 days post-operatively.
Myocardial Infarction (MI) | Within 30 days post-operatively
  Occurrence of Myocardial Infarction within 30 days post-operatively.
Cerebral Vascular Event (CVA) | Within 30 days post-operatively
  Occurrence of Myocardial Infarction within 30 days post-operatively.
Venous Thromboembolism (VTE) | Within 30 days post-operatively
  Occurrence of Venous Thromboembolism within 30 days post-operatively.
Acute Renal Failure (ARF) | Within 30 days post-operatively
  Occurrence of Acute Renal Failure within 30 days post-operatively.
Sepsis or septic shock | Within 30 days post-operatively
  Occurrence of sepsis or septic shock within 30 days post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Janny Xue Chen Ke, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris MS, Deierhoi RJ, Richman JS, Altom LK, Hawn MT. The relationship between timing of surgical complications and hospital readmission. JAMA Surg. 2014 Apr;149(4):348-54. doi: 10.1001/jamasurg.2013.4064. PMID 24522747
- [Background] Scarborough JE, Schumacher J, Kent KC, Heise CP, Greenberg CC. Associations of Specific Postoperative Complications With Outcomes After Elective Colon Resection: A Procedure-Targeted Approach Toward Surgical Quality Improvement. JAMA Surg. 2017 Feb 15;152(2):e164681. doi: 10.1001/jamasurg.2016.4681. Epub 2017 Feb 15. PMID 27926773
- [Background] Thompson JS, Baxter BT, Allison JG, Johnson FE, Lee KK, Park WY. Temporal patterns of postoperative complications. Arch Surg. 2003 Jun;138(6):596-602; discussion 602-3. doi: 10.1001/archsurg.138.6.596. PMID 12799329
- [Background] Luo W, Phung D, Tran T, Gupta S, Rana S, Karmakar C, Shilton A, Yearwood J, Dimitrova N, Ho TB, Venkatesh S, Berk M. Guidelines for Developing and Reporting Machine Learning Predictive Models in Biomedical Research: A Multidisciplinary View. J Med Internet Res. 2016 Dec 16;18(12):e323. doi: 10.2196/jmir.5870. PMID 27986644
- [Background] Riley RD, Snell KI, Ensor J, Burke DL, Harrell FE Jr, Moons KG, Collins GS. Minimum sample size for developing a multivariable prediction model: PART II - binary and time-to-event outcomes. Stat Med. 2019 Mar 30;38(7):1276-1296. doi: 10.1002/sim.7992. Epub 2018 Oct 24. PMID 30357870
- [Derived] Ke JXC, Jen TTH, Gao S, Ngo L, Wu L, Flexman AM, Schwarz SKW, Brown CJ, Gorges M. Development and internal validation of time-to-event risk prediction models for major medical complications within 30 days after elective colectomy. PLoS One. 2024 Dec 2;19(12):e0314526. doi: 10.1371/journal.pone.0314526. eCollection 2024. PMID 39621640

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT05150548/Prot_SAP_000.pdf